CLINICAL TRIAL: NCT06577480
Title: Investigation of Validity and Reliability of the Turkish Version of the Post-Liver Transplant Quality of Life (pLTQ) Questionnaire
Brief Title: Validity and Reliability of the Turkish Version of the Post-Liver Transplant Quality of Life Questionnaire
Status: Active, not recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak, Aslihan Cakmak-Onal, Hacettepe University
Other Study IDs: SBA 24/665
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Liver Transplant Disorder; Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplant recipients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Liver transplantation is a crucial treatment for life-threatening liver diseases, including acute liver failure, end-stage chronic liver disease, primary liver cancers, and congenital metabolic disorders. Quality of life in liver transplant patients is vital. The World Health Organization defines quality of life as an individual's perception of their position in life within the context of culture, values, goals, and expectations. Liver transplantation improves quality of life. Recipients should be closely monitored and supported psychologically, with the effectiveness of the intervention in improving quality of life well-documented. Saab et al. developed the post-Liver Transplantation Quality of Life (pLTQ) questionnaire, which includes eight sub-dimensions across 32 items. To our knowledge, no Turkish-specific QoL tool for liver transplant patients currently exists. This study aims to validate and assess the reliability of the Turkish version of the pLTQ questionnaire.

ELIGIBILITY:
Inclusion criteria:

* Being 18 years of age or older,
* Having received post-liver transplant treatment at Hacettepe University Adult Hospital General Surgery Units and being referred to Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit after routine clinical and laboratory examinations, if deemed appropriate for the study,
* Being willing to participate in the study.

Exclusion criteria:

* Having undergone combined liver-kidney transplantation and multiple organ transplantation,
* Having uncontrolled cardiovascular and neurological problems,
* Having a cognitive problem that will prevent understanding the questionnaires,
* Not being willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant recipients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Assessment of quality of life - disease specific | 1st day
  The post-Liver Transplant Quality of Life questionnaire consists of 32 items that assess specific factors that may affect the lives of liver transplant recipients, including symptoms, mood, limitation of activities of daily living, energy level, and transplant-related care. The items are scored on a seven-point Likert-type scale, where 1 means "always" and 7 means "never." Each subsection score and a total score are obtained with the post-Liver Transplant Quality of Life questionnaire. Higher values indicate higher quality of life.
Assessment of quality of life - general | 1st day
  In order to evaluate the validity of the Turkish post-Liver Transplant Quality of Life questionnaire, the Short Form-36 will be used. The Short Form-36 consists of eight sub-sections: physical function, social function, role restriction due to physical problems, role restriction due to emotional problems, mental health, vitality, body pain, general health, and change in health. Each sub-score is scored between 0 and 100. Higher scores indicate better quality of life.
Assessment of health profile | 1st day
  In order to evaluate the validity of the Turkish post-Liver Transplant Quality of Life questionnaire, Nottingham Health Profile will be used. Nottingham Health Profile consists of 38 items. It has six sub-sections: energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), and physical mobility (8 items). There is a possible score range for each sub-section ranging from 0 to 100 points. Higher scores indicate greater limitations in quality of life.
Psychosocial status assessment | 1st day
  The Hospital Anxiety and Depression Scale will be used to assess the anxiety and depression levels of patients. This scale consists of 14 items that aim to determine the risk of anxiety and depression in the patient, and to measure its level and severity change. The scale, which is asked to be answered by taking into account the last few days, has two subscales consisting of seven separate items measuring anxiety and depression. Higher scores indicate a better psychosocial status.
Fatigue assessment | 1st day
  The Fatigue Severity Scale will be used to assess fatigue. This scale questions the patient's fatigue status in the last month. The scale, which consists of a total of 9 items, is scored on a 7-point Likert type. The total score is calculated by taking the average of the items. As the score increases, the patient's perception of fatigue increases.

SECONDARY OUTCOMES:
Anthropometric and clinical characteristics | 1st day
  Demographic and anthropometric data of the patients, etiology of the disease (HCV, HBV, alpha-1 antitrypsin deficiency, hepatosteatosis, HCC, HCC+HBV, cryptogenic, ethanol, autoimmune hepatitis, etc.), duration of the disease and waiting times on the transplant list, medications used, other accompanying problems, donor characteristics will be questioned and data on laboratory tests will be recorded from the patient files. Risk factors such as smoking and alcohol use history, hypertension, diabetes mellitus will be questioned.
Model for End-Stage Liver Disease score index | 1st day
  Model for End-Stage Liver Disease score index will be used to determine the severity of chronic liver disease and it will be calculated with creatinine, bilirubin, international normalized ratio (INR), sodium and albumin values routinely checked in end-stage liver patients (https://medcalculators.stanford.edu/meld).

CONTACTS AND LOCATIONS:
Overall Officials: Aslihan Cakmak-Onal, PhD, PT, Principal Investigator — Hacettepe University; Naciye Vardar-Yagli, PhD, PT, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahmud N. Selection for Liver Transplantation: Indications and Evaluation. Curr Hepatol Rep. 2020;19(3):203-212. doi: 10.1007/s11901-020-00527-9. Epub 2020 Jun 19. PMID 32837824
- [Background] Akarsu M. Liver transplantation in Turkey: The importance of experience. Turk J Gastroenterol. 2018 Nov;29(6):629-630. doi: 10.5152/tjg.2018.81018. No abstract available. PMID 30381270
- [Background] Muller PC, Kabacam G, Vibert E, Germani G, Petrowsky H. Current status of liver transplantation in Europe. Int J Surg. 2020 Oct;82S:22-29. doi: 10.1016/j.ijsu.2020.05.062. Epub 2020 May 23. PMID 32454252
- [Background] Girgenti R, Tropea A, Buttafarro MA, Ragusa R, Ammirata M. Quality of Life in Liver Transplant Recipients: A Retrospective Study. Int J Environ Res Public Health. 2020 May 27;17(11):3809. doi: 10.3390/ijerph17113809. PMID 32471157
- [Background] Onghena L, Develtere W, Poppe C, Geerts A, Troisi R, Vanlander A, Berrevoet F, Rogiers X, Van Vlierberghe H, Verhelst X. Quality of life after liver transplantation: State of the art. World J Hepatol. 2016 Jun 28;8(18):749-56. doi: 10.4254/wjh.v8.i18.749. PMID 27366301
- [Background] Jay CL, Butt Z, Ladner DP, Skaro AI, Abecassis MM. A review of quality of life instruments used in liver transplantation. J Hepatol. 2009 Nov;51(5):949-59. doi: 10.1016/j.jhep.2009.07.010. Epub 2009 Jul 28. PMID 19775771
- [Background] Vedadi A, Khairalla R, Che A, Nagee A, Saqib M, Ayub A, Wasim A, Macanovic S, Orchanian-Cheff A, Selzner-Malekkiani N, Bartlett S, Mucsi I. Patient-reported outcomes and patient-reported outcome measures in liver transplantation: a scoping review. Qual Life Res. 2023 Sep;32(9):2435-2445. doi: 10.1007/s11136-023-03405-1. Epub 2023 Apr 6. PMID 37022585
- [Background] Rimmer B, Jenkins R, Russell S, Craig D, Sharp L, Exley C. Assessing quality of life in solid organ transplant recipients: A systematic review of the development, content, and quality of available condition- and transplant-specific patient-reported outcome measures. Transplant Rev (Orlando). 2024 Apr;38(2):100836. doi: 10.1016/j.trre.2024.100836. Epub 2024 Feb 13. PMID 38359538
- [Background] Saab S, Ng V, Landaverde C, Lee SJ, Comulada WS, Arevalo J, Durazo F, Han SH, Younossi Z, Busuttil RW. Development of a disease-specific questionnaire to measure health-related quality of life in liver transplant recipients. Liver Transpl. 2011 May;17(5):567-79. doi: 10.1002/lt.22267. PMID 21506245
- [Background] Kim WR, Mannalithara A, Heimbach JK, Kamath PS, Asrani SK, Biggins SW, Wood NL, Gentry SE, Kwong AJ. MELD 3.0: The Model for End-Stage Liver Disease Updated for the Modern Era. Gastroenterology. 2021 Dec;161(6):1887-1895.e4. doi: 10.1053/j.gastro.2021.08.050. Epub 2021 Sep 3. PMID 34481845
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Soyyigit S, Erk M, Guler N, Kilinc G. [The value of SF-36 questionnaire for the measurement of life quality in chronic obstructive pulmonary disease]. Tuberk Toraks. 2006;54(3):259-66. Turkish. PMID 17001544
- [Background] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- See also: Related Info — http://www.who.int/publications/i/item/WHO-HIS-HSI-Rev.2012.03
- See also: Related Info — http://dergipark.org.tr/tr/download/article-file/16232
- See also: Related Info — http://www.turkpsikiyatri.com/turkceOzet?Id=308
- See also: Related Info — http://jag.journalagent.com/kvhd/pdfs/KVHD-30164-RESEARCH_ARTICLE-SAYIN_KASAR.pdf